CLINICAL TRIAL: NCT03855267
Title: Effects of Etomidate/Propofol Mixture or Propofol Monotherapy With Different Proportions on Circulation and Prognosis in Patients Undergoing General Anesthesia
Brief Title: Etomidate/Propofol Mixture or Propofol Monotherapy Use in Patients Undergoing General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guolin Wang (Other)
Responsible Party: Sponsor-Investigator, Guolin Wang, Tianjin Medical University General Hospital, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GWang007
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Etomidate is Mixed With Propofol
Keywords: propofol; etomidate; General anesthesia; mixture
MeSH Terms: interventions — Propofol; Etomidate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Placebo Comparator): Propofol 20 mg/ml, recommended anesthesia induction dose of 0.1~0.125 ml/kg, anesthesia maintenance pump speed of 0.2~0.5ml/kg/h. keep bispectral index within 40 # 60
  Interventions: Drug: Propofol 20 MG/ML
- GroupB (Active Comparator): EP1:3, that is, 10ml etomidate was mixed with 30ml propofol, the recommended anesthesia induction dose was 0.1-0.125ml /kg, and the anesthesia maintenance pump speed was 0.2-0.5ml /kg/h.keep bispectral index within 40 # 60.Propofol 20 mg/ml,etomidate 2mg/ml.
  Interventions: Drug: Propofol 20 mg/ml , etomidate 2 mg/ml
- Group C (Active Comparator): EP1:1, that is, 20ml etomidate was mixed with 20ml propofol, the recommended anesthesia induction dose was 0.1-0.125ml /kg, and the anesthesia maintenance pump speed was 0.2-0.5ml /kg/h.keep bispectral index within 40 # 60.Propofol 20 mg/ml,etomidate 2mg/ml.
  Interventions: Drug: Propofol 20 mg/ml , etomidate 2 mg/ml
- Group D (Active Comparator): EP3:1, that is, 30ml etomidate was mixed with 10ml propofol, the recommended anesthesia induction dose was 0.1-0.125ml /kg, and the anesthesia maintenance pump speed was 0.2-0.5ml /kg/h.keep bispectral index within 40 # 60.Propofol 20 mg/ml,etomidate 2mg/ml.
  Interventions: Drug: Propofol 20 mg/ml , etomidate 2 mg/ml

INTERVENTIONS:
Drug: Propofol 20 MG/ML — Pump propofol to keep bispectral index within 40 # 60
  Arms: Group A
Drug: Propofol 20 mg/ml , etomidate 2 mg/ml — Propofol was mixed with etomidate in different proportions.keep bispectral index within 40 # 60.
  Arms: Group C; Group D; GroupB

SUMMARY:
The purpose of this study was to investigate the effects of different proportions of etomidate/propofol mixture and propofol alone intravenous anesthesia on intraoperative and postoperative physiological indicators and complications, and to find out the optimal use ratio of E/P mixture.

DETAILED DESCRIPTION:
Propofol is one of the most commonly used intravenous anesthesia drugs clinically, the pharmacokinetic characteristics makes it very suitable for total intravenous anesthesia( TIVA), etomidate belongs to intravenous anesthesia with propofol, is a derivative of the imidazoles, its calm performance is strong, work quickly, no obvious respiratory depression, had little effects on the cardiovascular system, which, therefore, to protect the cardiovascular, maintain hemodynamic stability has a certain advantage. Our previous project showed that propofol and etomidate combined application can maintain stable hemodynamics in patients with better, reduce the occurrence of adverse reactions, can be used within 3 h of surgery anesthesia.The purpose of this study is to use propofol or etomidate/propofol mixture in combination with BIS monitoring to perform general anesthesia maintenance for patients, in order to ensure the appropriate depth of anesthesia, better maintain the hemodynamic stability of patients, reduce adverse reactions, and find the appropriate E/P mixture of the best proportion and dose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective general anesthesia surgery in 3h;
2. American Society of Anesthesiologists gradesⅠ~III;
3. Aged 18 to 65 years, Body Mass Index 18.5 ~ 29.9kg / m2;
4. Hemoglobin 100 ~ 125g / L.
5. In line with the ethics, the patients volunteered to take the test and signed the informed consent

Exclusion Criteria:

1. Identify or suspect abuse or chronic use of narcotic sedatives and analgesics;
2. Heart, or liver, or lung, or kidney dysfunction;
3. Body mass index> 30kg / m2; or <18.5kg / m2
4. Speech, hearing or mental disorders;
5. severe diabetes, hyperkalemia ;
6. participate in other drug clinical researches in four weeks;
7. Poor compliance, can not complete clinical research by research program.
8. Any cerebrovascular accident occurred within 3 months, such as stroke, TIA, etc
9. Unstable angina and myocardial infarction occurred within 3 months;
10. Having contraindications or allergies to experimental drugs and other narcotic drugs;
11. Mental illness, hyperkalemia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
blood pressure | intraoperative
  the blood pressure is recorded (mmHg)
heart rate | intraoperative
  the heart rate is recorded(bpm)

SECONDARY OUTCOMES:
Perioperative complications | intraoperative
  the incidence of injection pain #nausea and vomit#intraoperative awareness and postoperative agitation.

OTHER OUTCOMES:
Recovery time | intraoperative
  Anesthesia awakening time and extubation time

CONTACTS AND LOCATIONS:
Overall Officials: Guolin Wang, MD.PHD, Study Director — Tainjin Medical University General Hospita
Locations (1):
- Zicheng Wang, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided